CLINICAL TRIAL: NCT02266407
Title: The Surgical and Economic Effect of the Aquamantys System in Blood Management During and Following Aseptic and Septic Revision TKA
Brief Title: Surgical / Economic Effect of the Aquamantys System in Blood Management for Aseptic and Septic Revision TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Surgical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TD-07711
Record Dates: First submitted 2012-10-19; First posted 2014-10-17 (Estimated); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Infection of Total Knee Joint Prosthesis; Aseptic Loosening of Prosthetic Joint
Keywords: Revision TKA; Septic; Aseptic; Transfusion; Blood Loss
MeSH Terms: conditions — Infertility; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ASEPTIC Revision TKA & Aquamantys System (Active Comparator): Single-stage revision TKA cases performed for aseptic failure requiring an extended osteotomy for component removal and intra-operative blood management (bipolar sealing) with the Aquamantys® System. These will be compared to in-house matched historic control using patients presenting with ASEPTIC failed primary TKA and revised without use of the Aquamantys® System.
  Interventions: Procedure: Aquamantys System
- SEPTIC Revision TKA & Aquamantys System (Active Comparator): Single-stage revision TKA cases performed for septic failure requiring an extended osteotomy for component removal and intra-operative blood management (bipolar sealing) with the Aquamantys® System. These will be compared to in-house matched historic control using patients presenting with SEPTIC failed primary TKA revised without use of the Aquamantys® System.
  Interventions: Procedure: Aquamantys System

INTERVENTIONS:
Procedure: Aquamantys System — The use of the saline-coupled bipolar sealing technology (Aquamantys® System, Medtronic Advanced Energy, LLC, Portsmouth, NH, USA) uses bipolar radiofrequency energy combined with a continuous-flow saline at the electrode tip to prevent tissue temperatures from exceeding 100 °C thus minimizing tissue charring. The temperature achieved is sufficient to induce a process called Transcollation(TM) which shrinks the collagen fibers in the walls of blood vessels, effectively sealing the blood vessels up to 1mm in diameter, resulting in the reduction of bleeding from soft tissue.

SUMMARY:
To assess the surgical and economic effectiveness of the Aquamantys System in managing intra- and post-operative blood loss, and reducing transfusion needs in patients undergoing both aseptic and septic revision total knee arthroplasty.

DETAILED DESCRIPTION:
The use of the saline-coupled bipolar sealing technology (Aquamantys® System, Medtronic Advanced Energy, LLC, Portsmouth, NH, USA) represents a modern approach to reducing perioperative blood loss in patients undergoing total joint arthroplasty. Unlike standard electrocautery, which use monopolar radiofrequency energy, this technology uses bipolar radiofrequency energy combined with a continuous-flow saline at the electrode tip to prevent tissue temperatures from exceeding 100 °C thus minimizing tissue charring. This eliminates the smoke and eschar formation seen with standard electrocautery. The temperature achieved is sufficient to induce a process called Transcollation(TM) which shrinks the collagen fibers in the walls of blood vessels, effectively sealing the blood vessels up to 1mm in diameter, resulting in the reduction of bleeding from soft tissue.

Suction is used to remove the saline from the surgical field with the treated tissue turning a light tan color. With normal use, the depth of penetration of this effect is typically less than 2mm. The technology is cleared by the US FDA (510(k)) and EU (CE Mark) for use on soft tissue & bone and will be used according to its intended packaging indications for use. The current assessment proposes a technique in which a disposable Aquamantys® hand piece is used to treat targeted areas which are bleeding or expected to bleed during surgery.

This postmarket study will assess the surgical and economic effectiveness of Aquamantys® System in managing intra-operative blood loss and transfusion rates in patients undergoing septic and aseptic revision TKA.

ELIGIBILITY:
Inclusion Criteria

* The patient is greater than 18 years of age
* Patients following failure of primary, unilateral TKA
* The degree of revision requires the use of an extended osteotomy for component removal
* Patient has participated in the informed consent process and has signed an Ethics Committee approved informed consent

Exclusion Criteria

* Patients presenting with a history of bleeding disorders and/or are on chronic blood anticoagulation therapy
* Patients presenting with an internal cardiac defibrillator
* Women who are pregnant
* Prisoner or transient
* Recent history of known narcotic abuse
* Any significant psychological disturbance past or present, that could impair the consent process or ability to complete subject self-report questionnaires
* Subject unwilling to undergo blood transfusion, if necessary

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Blood Loss and Post-Operative Transfusion Rate | 14 days
  To reduce blood loss and post-operative transfusion rates in patients undergoing total joint arthroplasty. This will be achieved using the Aquamantys system. The Aquamantys system provides transcollation which shrinks the collagen fibers in the walls of blood vessels, effectively sealing the blood vessels up to 1mm in diameter, resulting in the reduction of bleeding from soft tissue.

SECONDARY OUTCOMES:
Operative room and total hospital costs | 14 days
  The data to be collected will include, but is not limited to: copies of the subjects' hospital bills, corresponding Explanation of Benefits (EOB), physician's bill, or itemized hospital bills. The economic form(s) are collected and copies are provided to the sponsor.

OTHER OUTCOMES:
Change in hemoglobin and hematocrit from baseline (pre-op) | 14 days
  As data is collected from subject record an analysis of this data will provide changes in hemoglobin levels

CONTACTS AND LOCATIONS:
Overall Officials: Palaniswamy Vijay, PhD, Study Director — Medtronic Surgical Technologies; Joachim Singer, Dr.med., Principal Investigator — Orthopädische Klinik Markgröningen gGmbH
Locations (1):
- Orthopädische Klinik Markgröningen gGmbH, Markgröningen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bierbaum BE, Callaghan JJ, Galante JO, Rubash HE, Tooms RE, Welch RB. An analysis of blood management in patients having a total hip or knee arthroplasty. J Bone Joint Surg Am. 1999 Jan;81(1):2-10. doi: 10.2106/00004623-199901000-00002. PMID 9973048
- [Background] Marulanda GA, Krebs VE, Bierbaum BE, Goldberg VM, Ries M, Ulrich SD, Seyler TM, Mont MA. Hemostasis using a bipolar sealer in primary unilateral total knee arthroplasty. Am J Orthop (Belle Mead NJ). 2009 Dec;38(12):E179-83. PMID 20145794
- [Background] Marulanda GA, Ragland PS, Seyler TM, Mont MA. Reductions in blood loss with use of a bipolar sealer for hemostasis in primary total knee arthroplasty. Surg Technol Int. 2005;14:281-6. PMID 16525984
- [Background] Pfeiffer M, Brautigam H, Draws D, Sigg A. A new bipolar blood sealing system embedded in perioperative strategies vs. a conventional regimen for total knee arthroplasty: results of a matched-pair study. Ger Med Sci. 2005 Dec 13;3:Doc10. PMID 19675727
- [Background] Rosenberg AG. Reducing blood loss in total joint surgery with a saline-coupled bipolar sealing technology. J Arthroplasty. 2007 Jun;22(4 Suppl 1):82-5. doi: 10.1016/j.arth.2007.02.018. PMID 17570284